CLINICAL TRIAL: NCT00136513
Title: A Phase I Study to Determine the Safety and Pharmacokinetics of Intravenous Administration of SB743921 on a Once Every 3 Week Schedule in Patients With Solid Tumors
Brief Title: SB-743921 In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 743921/001
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Solid Tumor Cancer
Keywords: Safety; tolerability; dose limiting toxicity; solid tumors
MeSH Terms: interventions — SB 743921

INTERVENTIONS:
Drug: SB-743921

SUMMARY:
The purpose of this study is to find a dose of SB-743921 in adult patients with solid tumors or lymphoma who have progressed on standard therapy or who have relapsed. SB-743921 is dosed by 1-hour intravenous infusion every 3 weeks. A patient may continue to receive treatment as long as they are benefiting from the treatment. Blood samples will be taken at specific times to measure the amount of the drug in your body at specific times after the drug is given. Blood samples will also be taken for lab tests such as complete blood counts and clinical chemistries. Physical exams will be performed before each treatment with SB-743921. During the treatment phase, the patients will undergo regular assessments for safety and clinical response.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of: a) Advanced solid tumor malignancy that is not responsive to standard therapies or for which there is no standard therapy; OR b) B-cell or T-cell lymphoma (excluding HIV-associated lymphoma) that has relapsed or is refractory after prior chemotherapy or radiotherapy and autologous or allogeneic bone marrow transplantation (if appropriate) AND/OR for which salvage chemotherapy, radiotherapy, or bone marrow transplantation is not indicated or has been refused by the patient.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2.

Exclusion criteria:

* Pre-existing hemolytic anemia.
* Pre-existing peripheral neuropathy greater than or equal grade 2.
* Absolute neutrophil count less than 1,500/mm3.
* Platelets less than 100,000/mm3.
* Hemoglobin less than 9 g/dL.
* Total bilirubin greater than1.5 mg/dL.
* AST/ALT greater than 2.5 X upper limit of normal.
* Creatinine clearance less than or equal to 60 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-04

PRIMARY OUTCOMES:
Safety and tolerability will include evaluation of adverse events (AE) and changes from baseline in vital signs and clinical laboratory parameters. PK endpoints will include Cl, Vd, AUC, Cmax, and t½.

SECONDARY OUTCOMES:
Tumor response Comparison of pre and post-dose biomarker levels and/or correlation of pre-dose biomarker levels to any subsequent tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Madison, Wisconsin